CLINICAL TRIAL: NCT06883877
Title: The Effect of a Multi-modal Program on Fear of Cancer Recurrence, Breast Cancer Symptoms and Social Support in Breast Cancer Patients
Brief Title: The Effect of a Multi-modal Program on Fear of Cancer Recurrence in Breast Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LIU WEIMIN (Other)
Responsible Party: Sponsor-Investigator, LIU WEIMIN, Phd, Beijing Shijitan Hospital, Capital Medical University
Organization: Beijing Shijitan Hospital, Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IIT2024-135-003
Record Dates: First submitted 2025-03-09; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: fear of cancer recurrence; symptoms; social support
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-Modal Program (MMP) (Experimental): MMP includes three modules: addressing psychological problems such as FCR; addressing problems related to breast cancer symptoms; and addressing tangible problems such as social support. Each module is divided into the chemotherapy period (hospitalization) and the chemotherapy interval (post-discharge). Each phase involves face-to-face, digital, and remote tools, with the intervention lasting 8 weeks. Each module has a different goal, and depending on the goal setting, the topic of the intervention is different. The goal of the information education stage is to improve patients' overall understanding of the disease and pay attention to the psychological problems of FCR. The goal of coping skills is that through the practice of coping skills, patients can learn to change thoughts, problem emotions, and behaviors. The objective of social support group interaction is to strengthen their social support networks.
  Interventions: Other: Multi-Modal Program (MMP)
- Routine care (Other)
  Interventions: Other: Routine care

INTERVENTIONS:
Other: Multi-Modal Program (MMP) — MMP includes three modules: addressing psychological problems such as FCR; addressing problems related to breast cancer symptoms; and addressing tangible problems such as social support. Each module is divided into the chemotherapy period (hospitalization) and the chemotherapy interval (post-discharge). Each phase involves face-to-face, digital, and remote tools, with the intervention lasting 8 weeks. Each module has a different goal, and depending on the goal setting, the topic of the intervention is different. The goal of the information education stage is to improve patients' overall understanding of the disease and pay attention to the psychological problems of FCR. The goal of coping skills is that through the practice of coping skills, patients can learn to change thoughts, problem emotions, and behaviors. The objective of social support group interaction is to strengthen their social support networks.
  Arms: Multi-Modal Program (MMP)
Other: Routine care — The control group will receive routine care.
  Arms: Routine care

SUMMARY:
The goal of this clinical trial is to learn if MMP intervention can alleviate FCR , breast cancer symptoms and social support among breast cancer patients. he main questions it aims to answer are:

* Null Hypotheses (H0): There is no significant difference in FCR, breast cancer symptoms, and social support between the MMP intervention group and the control group.
* Alternative Hypotheses (H1): There are significant differences in FCR, breast cancer symptoms, and social support between the MMP intervention group and the control group

Researchers will compare MMP to a routine care to see if MMP works to alleviate FCR, breast cancer symptoms and social support.

Participants will:

* Receive interventions once per chemotherapy cycle for 8 weeks.
* The FCRI-SF, MSAS-SF-SC, and SSRS scales will be utilized to assess FCR levels, breast cancer symptoms and social support in both the experimental and control groups, with measurements conducted at baseline (T1), 8 weeks post-intervention (T2), and 12 weeks post-intervention (T3).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis meets the criteria outlined in the Breast Cancer Diagnosis and Treatment Guidelines, with a pathological diagnosis of breast cancer and currently undergoing chemotherapy
* Age ≥ 18 years
* Clear consciousness and the ability to communicate independently
* Aware of the diagnosis and has signed the informed consent form

Exclusion Criteria:

* Presence of mental illness or cognitive impairment
* Hearing or speech impairmen
* Distant metastasis of cance
* Severe physical illness or other malignant tumors requiring treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence Inventory-Short Form | baseline; 8 weeks post-intervention; 12 weeks post-intervention
  It consists of nine items, each of which is assessed using a 5-point Likert scale ranging from 0 to 4. The total score ranges from 0-36, with elevated scores reflecting heightened FCR
The Social Support Rating Scale | baseline; 8 weeks post-intervention; 12 weeks post-intervention
  This instrument comprises 10 items categorized into three dimensions, yielding a total score between 0 and 66, where elevated scores denote greater social support.
The Chinese version of memorial symptom assessment scal | baseline; 8 weeks post-intervention; 12 weeks post-intervention
  The scoring range for physical symptoms is from 0-4, whereas other items are scored from 1-4. Higher scores indicate greater distress.

IPD SHARING:
Plan to Share IPD: No